CLINICAL TRIAL: NCT02021461
Title: Double-blind Study in Paediatric Epileptic Subjects Aged From 5 to Less Than 8 Years to Compare the Subject Preference for ESL Suspension Formulation With Alternative Flavours
Brief Title: Double-blind Study in Paediatric Epileptic to Compare the Subject Preference for ESL Suspension Formulation With Alternative Flavours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: BIA-2093-212
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ESL Banana taste (Experimental): Subjects were to be enrolled until there were at least 30 evaluable subjects (of whom at least 60% were <7 years of age). Evaluable subjects were those who completed 3 Visual analogue scale (VAS), 1 for each of the 3 tasting steps with the 3 flavoured oral suspensions.
  Interventions: Drug: ESL Banana taste
- ESL Grape taste (Experimental): Subjects were to be enrolled until there were at least 30 evaluable subjects (of whom at least 60% were <7 years of age). Evaluable subjects were those who completed 3 Visual analogue scale (VAS), 1 for each of the 3 tasting steps with the 3 flavoured oral suspensions.
  Interventions: Drug: ESL Grape taste
- ESL Tutti-Frutti taste (Experimental): Subjects were to be enrolled until there were at least 30 evaluable subjects (of whom at least 60% were <7 years of age). Evaluable subjects were those who completed 3 Visual analogue scale (VAS), 1 for each of the 3 tasting steps with the 3 flavoured oral suspensions.
  Interventions: Drug: ESL Tutti-Frutti taste

INTERVENTIONS:
Drug: ESL Banana taste — oral suspension with Banana flavor at a concentration of 50 mg/mL and was administered in 2.5 mL doses.
  Other Names: Eslicarbazepine acetate (ESL)
  Arms: ESL Banana taste
Drug: ESL Grape taste — oral suspension with Grape flavor at a concentration of 50 mg/mL and was administered in 2.5 mL doses.
  Other Names: Eslicarbazepine acetate (ESL)
  Arms: ESL Grape taste
Drug: ESL Tutti-Frutti taste — oral suspension with Tutti-Frutti flavor at a concentration of 50 mg/mL and was administered in 2.5 mL doses.
  Other Names: Eslicarbazepine acetate (ESL)
  Arms: ESL Tutti-Frutti taste

SUMMARY:
The purpose of this study is to investigate the taste preference in children of 3 different flavours of the ESL oral suspension.

DETAILED DESCRIPTION:
Children between the age of 5 and <8 years who are patients of the participating investigators will be screened for participation in the study. This may be at a regularly planned visit or the investigators may invite children who would be suitable candidates. Children who agree to participate will be invited to come back to the clinic on a single Study Day and will be randomised to a particular sequence of flavours. On the Study Day, all children will be given 3 different flavoured samples of Eslicarbazepine acetate (ESL) oral suspension for tasting, in the sequence to which they were randomised, in a double-blind, standardized setting. Each sample will consist of 2.5 mL and is to be given with a spoon in a double-blind manner, and is not to be swallowed. After tasting and spitting out each sample the child will be asked to rate the taste on a 10 cm visual analogue scale incorporating a facial hedonic scale. At the end of the session, the child will also be asked which flavour they thought tasted the best and which tasted the worst, to assess overall taste. A follow-up telephone contact interview will be performed between 1 and 4 days after the Study Day to collect adverse event (AE) data.

ELIGIBILITY:
Inclusion Criteria:

* A written informed consent form signed by the subject's parent(s) or guardian(s) and an assent form for any 7-year-old subjects signed by subjects.
* Male or female, between the age of 5 to <8 years.
* Diagnosed with partial-onset epilepsy.
* Is considered, in the opinion of the investigator, to be able to make the required taste assessment.

Exclusion Criteria:

* Uncontrolled cardiac, renal, hepatic, endocrine, gastrointestinal, metabolic, haematological, or oncology disorder.
* Known hypersensitivity to carboxamide derivatives or tricyclic antidepressants.
* Strong congestion, flu, or any other acute illness that could influence the child's sense of taste.
* A known swallowing or taste perception problem.
* Currently or previously treated with ESL.
* Concomitant participation in another drug clinical trial.
* Any other condition or circumstance that, in the opinion of the investigator, could compromise the subject's ability to comply with the study protocol.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Romania (2):
  - Dr. Bacos Cosma Medical Centre, Timișoara, Timiș County
  - Psychiatry Clinical Hospital "Prof. Dr. Alexandru Obregia" - Department of Pediatric, Bucharest
- Neurology Outpatient Clinic for children and adults, Bardejov, Slovakia

RESULTS

PARTICIPANT FLOW:
Groups:
- Eslicarbazepine Acetate: Eslicarbazepine acetate (ESL) was supplied as an oral suspension with 3 different flavours at a concentration of 50 mg/mL and was administered in 2.5 mL doses.
Period: Overall Study
Arm/Group | Eslicarbazepine Acetate
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 38 subjects were screened. All of these subjects were randomised and completed the trial
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Taste Preference
Description: Subject preference for 3 flavours of the ESL oral suspension was assessed based on a measured score using a 0-10 cm (minimum and maximum measured values) Visual Analogue Scale (VAS). Higher values represent the stronger preference.
Time Frame: single Study Day
Measure: Mean (Standard Deviation); unit: units on a scale (0-10 cm VAS)
Groups:
- ESL Banana Taste: ESL was supplied as an oral suspension with 3 different flavours at a concentration of 50 mg/mL and was administered in 2.5 mL doses.
  ESL Banana taste
- ESL Grape Taste: ESL was supplied as an oral suspension with 3 different flavours at a concentration of 50 mg/mL and was administered in 2.5 mL doses.
  ESL Grape taste
- ESL Tutti-Frutti Taste: ESL was supplied as an oral suspension with 3 different flavours at a concentration of 50 mg/mL and was administered in 2.5 mL doses.
  ESL Tutti-Frutti taste
Arm/Group | ESL Banana Taste | ESL Grape Taste | ESL Tutti-Frutti Taste
Number analyzed (Participants) | 38 | 38 | 38
units on a scale (0-10 cm VAS) | 5.8 (3.5) | 5.8 (3.5) | 7.1 (3.2)

ADVERSE EVENTS:
Time Frame: After the first tasting of study treatment until 1-4 days after tasting the IMP
Description: The study comprised a Screening Visit (not more than 1 month before the Study Day), a single Study Day (which could occur on the same day as the Screening Visit), and a follow-up telephone contact interview (that was to be performed between 1 and 4 days after the Study Day). Thus, individual study durations may have been between 2-6 days.
Groups:
- Eslicarbazepine Acetate: Eslicarbazepine acetate (ESL) supplied as an oral suspension with 3 different flavours at a concentration of 50 mg/mL and was administered in 2.5 mL doses.
Arm/Group | Eslicarbazepine Acetate
Serious Adverse Events (participants affected / at risk) | 1/38
Other Adverse Events (participants affected / at risk) | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eslicarbazepine Acetate (N=38)
Laryngitis (Infections and infestations) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other